CLINICAL TRIAL: NCT05442645
Title: Observational Study of Atopic Dermatitis Patients Treated With Dupilumab in Taiwan
Brief Title: A Study in Male and Female Adult Patients With Atopic Dermatitis Treated With Dupilumab in Taiwan
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS17337; U1111-1269-6392 (Registry Identifier: ICTRP)
Record Dates: First submitted 2022-06-22; First posted 2022-07-05 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with AD: Male or female, 18 years or older at the baseline visit initiated treatment with dupilumab for AD, who are eligible for dupilumab reimbursement according to the country-specific prescribing information

SUMMARY:
Primary objective:

To characterize the use patterns of phototherapy and immunosuppressants prior to dupilumab treatment for adult AD patients, who are eligible for dupilumab reimbursement in Taiwan (e.g., used regimens, reason for initiation of new treatments, concomitant therapies, treatment durations and reasons for discontinuation and/or switching).

Secondary objectives:

* To characterize the adult AD patients, who are eligible for dupilumab reimbursement in Taiwan, with respect to their a) medical history, b) socio-demographic, c) disease characteristics, d) comorbid with type 2 diseases [e.g., Asthma, Chronic rhinosinusitis with nasal polyp (CRSwNP)], and e) prior and concomitant treatments of atopic dermatitis
* To assess the effectiveness and safety of dupilumab in adult atopic dermatitis patients, who are eligible for dupilumab reimbursement in Taiwan
* To assess comorbid atopic conditions and effects of dupilumab treatment for comorbid atopic conditions in adult patients, who are eligible for dupilumab reimbursement in Taiwan
* To evaluate the correlation of patient reported outcome [Atopic Dermatitis Control Tool (ADCT)] and physician assessment [Eczema Area and Severity Index (EASI)] from the recruited subjects

DETAILED DESCRIPTION:
1 year

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years or older at the baseline visit
* Initiating treatment with dupilumab for AD, who are eligible for dupilumab reimbursement according to the country-specific prescribing information

Note: Patients, who are diagnosed with AD more than 6 months, Eczema Area and Severity Index (EASI) more than or equals to 20. body surface area (of AD involvement) (BSA) more than or equals to 30% and IGA=3-4, may be eligible if they have already initiated treatment with:

1. Phototherapy (psoralen + ultraviolet light A (PUVA) or narrow-band ultraviolet B (nb-UVB) twice a week) more than 3 months, and,
2. Two different immunosuppressants (methotrexate, azathioprine, or cyclosporine) more than 3 months respectively before their enrollment in the registry.

   * Provided signed informed consent

Exclusion Criteria:

* Any condition that, in the opinion of the Investigator, may interfere with patient's ability to participate in the study, such as short life expectancy, substance abuse, severe cognitive impairment, or other comorbidities that can predictably prevent the patient from adequately completing the schedule of visits and assessments
* Patients currently participating in any interventional clinical trial which modifies patient care
* Patients who have a contraindication to dupilumab according to the country-specific prescribing information

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AD patients, who are eligible for dupilumab reimbursement in Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Characterization of the use patterns of phototherapy and immunosuppressants prior to dupilumab treatment: Used regimens | At baseline (Day 1)
Characterization of the use patterns of phototherapy and immunosuppressants prior to dupilumab treatment: Reason for initiation of new treatments | At baseline (Day 1)
Characterization of the use patterns of phototherapy and immunosuppressants prior to dupilumab treatment: Concomitant therapies | At baseline (Day 1)
Characterization of the use patterns of phototherapy and immunosuppressants prior to dupilumab treatment: Treatment durations | At baseline (Day 1)
Characterization of the use patterns of phototherapy and immunosuppressants prior to dupilumab treatment: Reasons for discontinuation and/or switching | At baseline (Day 1)

SECONDARY OUTCOMES:
Characterization of the patients who receive dupilumab for AD: Medical history | At baseline (Day 1)
Characterization of the patients who receive dupilumab for AD: Socio-demographic data | At baseline (Day 1)
Characterization of the patients who receive dupilumab for AD: Prior and concomitant treatments of AD; percentage who were on dupilumab at the baseline/enrollment visit (Visit 1) | At baseline (Day 1)
Characterization of the patients who receive dupilumab for AD: Reason for initiation of dupilumab | At baseline (Day 1)
Characterization of the patients who receive dupilumab for AD: Baseline assessments of comorbid conditions (Asthma Control Questionnaire (ACQ-5)) | At baseline (Day 1)
Characterization of the patients who receive dupilumab for AD: Baseline assessments of comorbid conditions (22-item Sino-Nasal Outcome Test (SNOT-22)) | At baseline (Day 1)
Characterization of real-world use patterns of dupilumab for AD: Dupilumab dose regimens used over the study, and the duration with each regimen | Up to 12 months
Characterization of real-world use patterns of dupilumab for AD: Percentage of patients whose dose (either the frequency of the strength) increased from starting regimen and reasons; percentage whose dose decreased from the starting regimen and reasons | Up to 12 months
Characterization of real-world use patterns of dupilumab for AD: Percent discontinuing dupilumab, including temporary or permanent discontinuation; reasons for discontinuation | Up to 12 months
Characterization of real-world use patterns of dupilumab for AD: Longest duration of use | Up to 12 months
Characterization of real-world use patterns of dupilumab for AD: Number of gaps in dupilumab treatment and longest gap length | Up to 12 months
Characterization of real-world use patterns of dupilumab for AD: Concomitant therapies taken for AD | Up to 12 months
Effectiveness of dupilumab: change from baseline in Eczema Area and Severity Index (EASI) | Day 0, Months 3, 6, 9 and 12
Effectiveness of dupilumab: change from baseline in body surface area (of AD involvement) (BSA) | Day 0, Months 3, 6, 9 and 12
Effectiveness of dupilumab: change from baseline in Investigator global assessment scale (IGA) | Day 0, Months 3, 6, 9 and 12
Effectiveness of dupilumab: change from baseline in Scoring of Atopic Dermatitis (SCORAD) | Day 0, Months 3, 6, 9 and 12
Effectiveness of dupilumab: change from baseline in Patient-Oriented Eczema Measure (POEM) | Day 0, Months 3, 6, 9 and 12
Effectiveness of dupilumab: change from baseline in Atopic Dermatitis Control Tools (ADCT) | Day 0, Months 3, 6, 9 and 12
Effectiveness of dupilumab: change from baseline in Pruritus Numerical Rating Scale (NRS) | Day 0, Months 3, 6, 9 and 12
Effectiveness of dupilumab: change from baseline in Sleep NRS | Day 0, Months 3, 6, 9 and 12
Effectiveness of dupilumab: change from baseline in Dermatology Life Quality Index (DLQI) | Day 0, Months 3, 6, 9 and 12
Effectiveness of dupilumab in relevant comorbid conditions: change in Juniper Asthma Control Questionnaire (ACQ-5) from the first reported time point of Asthma | Day 0 to Month 12
Effectiveness of dupilumab in relevant comorbid conditions: change in 22-item Sino-Nasal Outcome Test (SNOT-22) from the first reported time point of Asthma | Day 0 to Month 12
Percentage of participants reporting that their comorbid condition got better, and the percentage reporting their condition got worse at each follow-up visit by each specific condition (other than asthma and allergic rhinitis) | Day 0 to Month 12
Safety: Number of patients with at least 1 adverse event (AE) | Day 0 to Month 12
Safety: Annualized event rates of AEs | Day 0 to Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational site-National Taiwan University Hospital, Taipei, Taiwan, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org